CLINICAL TRIAL: NCT06034457
Title: 24 Week External Single-arm Study Testing the Effectiveness of WW GLP1 Behavioral Program + Sequence Medical Weight Management on Weight Loss and Related Outcomes
Brief Title: Testing the Effectiveness of WW Clinic GLP1
Acronym: WW Clinic
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, leslie heinberg, Professor, The Cleveland Clinic
Other Study IDs: 23-814
Record Dates: First submitted 2023-08-24; First posted 2023-09-13 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study objective is to evaluate the efficacy of the WeightWatchers (WW) GLP-1 behavioral program + WW Clinic (formerly known as Sequence medical weight management program) on weight loss and related outcomes. Participants will be invited to take part and answer surveys at 0, 12 and 24 weeks.

DETAILED DESCRIPTION:
This is a 24 week prospective single-arm efficacy outcomes study. Up to 180 adult participants who are currently enrolled in WW GLP-1 behavioral program program + WW Clinic (formerly known as Sequence medical weight management program) and already prescribed semaglutide or tirzepatide. The application of a comprehensive lifestyle-based intervention focused on dietary intake, physical activity, support and behavioral principles in conjunction with anti-obesity medication (AOM) is novel and may increase AOM efficacy while minimizing maintenance concerns. As obesity care can now be delivered virtually, it will also include an innovative strategy of virtual/remotely delivered medical care via Sequence and WW. Further, this study will examine multiple psychosocial domains associated with weight loss and weight loss related outcomes including physical activity, dietary behavior, disordered eating, depression symptoms, internalized weight bias and community, that have not been examined in AOM trials.

ELIGIBILITY:
Inclusion criteria:

1. 18 years or older
2. BMI of >30 or BMI of >27 with one or more weight related medically qualifying condition (hypertension, dyslipidemia, sleep apnea, cardiovascular disease)
3. Access to a smartphone or tablet that runs iOS/iPadOS 15.0 or later, or Android 7.0 or later
4. A prescription for Wegovy, Mounjaro, or Zepbound

Exclusion criteria:

1. Diabetes
2. Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia type 2
3. History of pancreatitis within 180 days
4. Previous surgical obesity treatment
5. Use of other anti-obesity medication in last 90 days
6. Use of GLP-1 within the last 180 days
7. Lost weight >11 lbs in the last 90 days
8. Pregnant, breastfeeding, intends to become pregnant, of child-bearing potential and not using a highly effective contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who are already enrolled in WW Clinic (formerly known as Sequence) and prescribed GLP-1 medications.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy DiVita, Study Director — The Cleveland Clinic; Matthew Allman, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinberg LJ, Lee AM, Foster GD, DiVita A, Allman M, Rotroff D, Dargham CB, Cardel MI. Effectiveness of Telemedicine Prescribing and a Long-Acting Obesity Medication Behavioral Program: A 24-Week Single-Arm Study. Obesity (Silver Spring). 2025 Nov 18. doi: 10.1002/oby.70056. Online ahead of print. PMID 41253738

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: WW GLP-1 behavioral program program + Sequence medical weight management prescribed semaglutide or tirzepatide.
Period: Overall Study
Arm/Group | Single Arm
Started | 180
Completed | 166
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.11 (10.41)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 16
  Female | 164
  Intersex | 0
  Prefer not to say | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 166
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 20
  White | 146
  More than one race | 4
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight in Pounds From Week 0 to Week 24
Description: Effect of WW GLP1 behavioral program + WW Clinic (formerly known as Sequence) on absolute change of weight loss at 24 weeks.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Single Arm
Number analyzed (Participants) | 180
pounds | -27.41 (14.86)

2. Secondary Outcome: Weight Loss Percentage Change From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on weight loss and % reaching 5, 10, 15, 20 % body weight loss at 24 weeks.
Time Frame: 0 to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 180
Participants
  Number of participants with >= 5% weight loss at 24 weeks | 161
  Number of participants with >= 10% weight loss at 24 weeks | 121
  Number of participants with >= 15% weight loss at 24 weeks | 81
  Number of participants with >= 20% weight loss at 24 weeks | 20

3. Other Pre Specified Outcome: Blood Pressure Changes (Systolic and Diastolic) in mmHg From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of blood pressure at 24 weeks
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Arm
Number analyzed (Participants) | 180
mmHg
  Change in diastolic blood pressure at 24 weeks | -5.66 (13.29)
  Change in systolic blood pressure at 24 weeks | -11.17 (14.96)

4. Other Pre Specified Outcome: Change in Quality of Life Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Quality of Life (QOL) scores using "Impact of Weight on Quality of Life-Lite Scale" Scale Name + Description of scale: "Impact of Weight on Quality of Life-Lite (IWQOL-Lite) Is a validated, 31-item, self-report measure of obesity-specific quality of life in adults. There are five domains include physical function, self-esteem, sexual life, public distress and work.
  Scale Ranges (min, max): 0-100 Description of scoring: Higher scores represent lower quality of life (i.e., greater impact of obesity on quality of life). Lower scores represent a better quality of life (i.e., less impact of obesity). A negative mean change indicates improvement in quality of life.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale
  Physical Function | -20.13 (17.79)
  Self-Esteem | -27.98 (22.5)
  Sexual Life | -18.27 (23.1)
  Public Distress | -11.44 (17.99)
  Work | -12.08 (19.81)
  Total Score | -19.19 (13.42)

5. Other Pre Specified Outcome: Changes in Well-being Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Well-being at 24 weeks using "WHO Well-Being Index 5" Scale Name + Description of scale: "Well-being Index 5 (WHO-5)" is a 5-item questionnaire that assesses subjective well-being through five statements about feeling cheerful, calm, active, interested and rested over the past two weeks.
  Scale Ranges (min, max) 0-25 Description of scoring: Lower scores indicate worse overall well-being, higher scores indicate better overall well-being. A positive mean change indicates improvement in well-being.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | 2.92 (3.98)

6. Other Pre Specified Outcome: Changes in Disordered Eating Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Disordered Eating at 24 weeks using "Eating Disorder Examination-Questionnaire" Scale Name + Description of scale: "Eating Disorder Examination-Questionnaire (EDE-Q)" is a 28-item self-report questionnaire, adapted from the semi-structured interview, the Eating Disorder Examination (EDE). The questionnaire is designed to assess the range, frequency and severity of behaviors associated with a diagnosis of an eating disorder.
  Scale Ranges (min, max): 0-6 Description of scoring: Lower scores indicate less problematic eating disordered behaviors and cognitions and higher scores indicate more problematic eating disordered behaviors and cognitions. A positive mean change indicates an increase in eating disordered symptoms. A negative mean change could indicate a decrease in eating disorder symptoms.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale
  Restraint Score | 0.09 (1.74)
  Eating Concerns Score | -0.75 (1.28)
  Shape Concern Score | -1.04 (1.07)
  Weight Concern Score | -0.76 (0.8)
  Global Score | -0.61 (0.95)

7. Other Pre Specified Outcome: Changes in Strength Training Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Strength Training Behavior at 24 weeks using the "Strength Training Behavior Scale" Scale Name + Description of scale: "Stage of Change for Strength Training" Strength training is defined as all activities that serve to enhance muscle strength and endurance (free weights, body weight exercises, etc.) Regular resistance training is described as engaging in these activities at least two times per week.
  Scale Ranges (min, max): 0-7 Description of scoring: Lower scores indicate less days strength training. Higher scores equal more days of strength training. A positive mean change indicates an increase in number of days of strength training.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | 0.48 (1.37)

8. Other Pre Specified Outcome: Changes in Stress Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Stress at 24 weeks using the "Perceived Stress Scale" Scale Name + Description of scale: "Perceived Stress Scale, PSS-10" is a self-report scale that asks about feelings and thoughts related to stressful things during the last month.
  Scale Ranges (min, max): 10-50 Description of scoring: Higher scores indicate more perceived stress and lower scores indicate less perceived stress. A negative mean change indicates improvement in perceived stress.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | -2.66 (6.51)

9. Other Pre Specified Outcome: Changes in Emotional Eating Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Emotional Eating scores using the "Palatable Eating Motives Scale-Coping Subscale" Scale Name + Description of scale: "Palatable Eating Motives Scale - Coping Subscale (PEMs-Coping)" is a four-item coping subscale of the PEMs self-report that measures eating behavior as a method of coping with problems and negative feelings.
  Scale Ranges (min, max): 4-20 Description of scoring: Lower scores indicate lower frequency of eating as a method of coping with problems and negative feelings. Higher scores indicate higher frequency of eating as a method of coping with problems and negative feelings. A negative mean score indicates a decrease in using eating to cope with problems and negative feelings.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | -3.99 (4.79)

10. Other Pre Specified Outcome: Changes in UnHealthy Habits Strength Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Unhealthy Habits scores using "Self-Reported Behavioral Automaticity Index" Scale Name + Description of scale: "Self-Reported Behavioral Automaticity Index (SRBAI)-Unhealthy Habits Subscale" is a self-report measure to assess how automatic or habitual certain behaviors are, often used to understand unhealthy habits. Unhealthy habits included are eating sugary foods, fried foods and drinking sugary drinks.
  Scale Ranges (min, max): 1-7 Description of scoring: Lower scores indicate less automatic or habitual unhealthy habits. Higher scores indicate more automatic or habitual unhealthy habits. A negative mean change indicates a decrease in automatic or habitual unhealthy behaviors.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale
  Sugary Foods | -1.64 (1.86)
  Fried Foods | -1.13 (1.81)
  Drinking | -0.83 (1.66)

11. Other Pre Specified Outcome: Changes in Healthy Habits Strength Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Habit Strength scores using the "Self-Reported Behavioral Automaticity Index for Healthy Habits" Scale Name + Description of scale: "Self-Reported Behavioral Automaticity Index (SRBAI) Healthy Habits Subscale" is a self-report measure to assess how automatic or habitual certain behaviors are, often used to understand healthy habits. Healthy habits included are portion control, food tracking, protein content, eating vegetables, weighing self, physical activity, positive self-talk after a setback, arranging kitchen so healthy foods are easy to access and meal planning.
  Scale Ranges (min, max): 1-7 Description of scoring: Lower scores indicate less automatic or habitual healthy habits. Higher scores indicate more automatic or habitual healthy habits. A positive mean change indicates an increase in automatic or habitual healthy behaviors.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale
  Portion | 1.72 (1.68)
  Tracking | 0.55 (1.86)
  Points | 1.24 (1.82)
  Vegetables | 0.48 (1.4)
  Weighing | 1.29 (2.01)
  Physically | 1.02 (1.57)
  Self-Talk | 0.82 (1.74)
  Healthy Food | 0.97 (1.79)
  Snacking | 0.61 (1.81)

12. Other Pre Specified Outcome: Changes in Weight Bias Internalization Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Weight Bias Internalization scores using "Weight Bias Internalization Scale" Scale Name + Description of scale: "Weight Bias Internalization Scale, WBIS-2F" is a 13-item measure developed to assess weight related self-stigma.
  Scale Ranges (min, max): 13-91 Description of scoring: Lower scores indicate more weight related self-stigma, higher scores indicate less weight related self-stigma. A negative mean change indicates a decrease in weight related self-stigma.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | -7.12 (9.83)

13. Other Pre Specified Outcome: Changes in Self-Compassion Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Self-Compassion scores using the "Self-Compassion Scale" Scale Name + Description of scale: "Self-Compassion Scale" is a self-report questionnaire that asks how someone typically acts towards themselves in difficult times.
  Scale Ranges (min, max): 1-5 Description of scoring: Lower scores indicate that an individual might be more critical of themselves during difficult times. Higher scores might indicate someone who might be less critical on themselves during difficult times. A positive mean change indicates more self-compassion.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | 0.05 (0.32)

14. Other Pre Specified Outcome: Number of Participants With GLP1 Side Effects From Week 0 to Week 24
Description: Number of Participants with GLP1 Side Effects from week 0 to week 24
Time Frame: 0 to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 180
Participants
  Nausea | 146
  Other | 67
  Constipation | 54
  Diarrhea | 41
  Abdominal Pain | 13
  Complete Lack of Appetite | 10
  Injection Site Reaction | 7
  Hair Loss | 4

15. Other Pre Specified Outcome: Changes in Restraint/Disinhibition Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Restraint/Disinhibition scores using the "Three Factor Eating Questionnaire" Scale Name + Description of scale: "Three Factor Eating Questionnaires, TFEQ". Is a self-report scale that measures three dimensions of eating behavior: cognitive restraint, disinhibition and hunger. The first two factors were included.
  Scale Ranges (min, max): restraint 0-21, disinhibition 0-16 Description of scoring: Lower scores indicate less restraint. Higher scores indicate more restraint. A positive change indicates improvement in restraint. Lower scores indicate less disinhibition. Higher scores indicate more disinhibition. A negative mean change improvement in disinhibition.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale
  Restraint Score | 2.42 (4.03)
  Disinhibition Score | -3.72 (3.49)

16. Other Pre Specified Outcome: Changes in Depression Symptom Scores From Week 0 to Week 24
Description: Effect of WW + WW Clinic (formerly known as Sequence) on absolute change of Depression symptoms using the "Patient Health Questionnaire-8"
  Scale Name + Description of scale: "Patient Health Questionniare-8 item" is a self-report scale that rates depressive symptoms including questions about interest, enjoyment, sadness, sleep, appetite, energy, guilt, concentration.
  Scale Ranges (min, max): 0-24
  Description of scoring: Lower scores indicate fewer depressive symptoms, higher scores indicate more depressive symptoms. A negative mean change indicates an improvement in depressive symptoms.
Time Frame: 0 to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 180
score on a scale | -2.99 (4.59)

ADVERSE EVENTS:
Time Frame: Week 0 to Week 24
Description: There were no adverse events during the collection of this observational survey study. Side effects related to GLP1s were gathered and reported by WW but there were no adverse events during the conduct of this observational study.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180
Other Adverse Events (participants affected / at risk) | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT06034457/Prot_SAP_000.pdf